CLINICAL TRIAL: NCT03549091
Title: Accuracy of Left Subclavian Regurgitation Evaluated by Ultrasound Doppler and 4D Flow MRI as an Indicator of Severe Aortic Regurgitation
Brief Title: Accuracy of Left Subclavian Regurgitation Evaluated by Ultrasound Doppler and 4D Flow MRI
Acronym: SUBCLAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SUBCLAR
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transthoracic echocardiography and MRI (Experimental): The TransThoracic Echocardiography imaging data are collected exactly as for a standard examination. However, an additional measurement of the flow at the level of the left subclavian artery is performed, resulting in a 10-minute increase in the examination time. A Cardiovascular Magnetic Resonance Imaging 4D Flow is programmed within a maximum of 10 (no change in treatment that could skew the comparison). The usual procedure for MRI is not modified. The examination allows the acquisition of conventional 2D sequences of flow measurements, regurgitant volume and regurgitation fraction obtained at the level of the descending aorta and the sino-tubular junction of the ascending aorta. An additional 4D sequence is acquired increasing the examination time by 10 minutes.
  Interventions: Diagnostic Test: transthoracic echocardiography; Diagnostic Test: Cardiovascular Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: transthoracic echocardiography — This involves the acquisition of 1 additional sequence: a 10-minute sequence for transthoracic echocardiography.
Diagnostic Test: Cardiovascular Magnetic Resonance Imaging — This involves the acquisition of 1 additional sequence: a 10-minute sequence for Cardiovascular Magnetic Resonance Imaging 4D Flow.

SUMMARY:
Aortic insufficiency (IA) is defined as an abnormal regurgitation of blood from the aorta to the left ventricle in diastole, due to a lack of tightness of the aortic valves. It represents about 10% of valvular pathologies but the annual mortality of nonoperated patients can be as high as 10% to 20%. The quantification of AI is therefore important as it can remain perfectly asymptomatic for a long time.

Doppler echocardiography is currently the key examination to confirm the presence of valvulopathy, to allow positive diagnosis of valve leakage regardless of location, to specify the etiology and mechanism of regurgitation. The quantification of IA requires, in transthoracic ultrasound, to take into account many parameters that individually have all certain limitations. The recommendations are therefore to have an integrative approach considering a combination of different parameters and an overall interpretation. This makes it possible to evaluate with greater precision the importance of the leak. Thus, there is the difficulty of quantifying moderate and severe AI for lack of a truly unique criterion. One of the evaluation criteria commonly used in transthoracic ultrasound is diastolic regurgitation in the aortic arch but this assessment is sometimes difficult. The left subclavian artery (SCG) is more accessible than the aortic arch in terms of the ultrasound window. The measurements will be easier to record since the vessel is more superficial and there are fewer air interpositions than for the aortic arch. The quantification of the AI based on this new element will be compared to the other previously validated ultrasound criteria. The investigators will use this study to describe the feasibility of collecting coronary flow in the artery (IVA), and they will compare systolic velocity, diastolic rate / systolic rate ratio compared to a control group without severe aortic insufficiency (grades 2 and 3). The flows recorded in the IVA will be compared to the importance of the aortic leakage according to its different modes of quantification (ultrasound and MRI). The aim of the study will be to show that diastolic reflux in the left subclavian artery is a marker of severe AI (grades 2 and 3) by comparing this regurgitation with that measured at the level of the aortic arch and other validated ultrasound criteria and cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient able to give informed consent to participate in the study
* Patient with transthoracic echocardiography and MRI prescription

Exclusion Criteria:

* Contraindication to MRI
* Pathologies of the thoracic aorta (aneurism, dissection, stenosis)
* Pathologies of the left subclavian artery (stenosis, narrowing)
* Persistent arterial canal
* Arteriovenous fistula of the upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of absence of reflux in the left subclavian artery in transthoracic echocardiography and MRI 4D flow | Day 1
  It allows to evaluate the sensitivity/specificity of the presence of the left subclavian artery based holodiastolic regurgitation using transthoracic echocardiography on the one hand and 4D flow MRI on the other hand compared to the validated combined sonographic quantification criteria.

SECONDARY OUTCOMES:
Establish a tele-diastolic velocity threshold at the level of the left subclavian artery to quantify aortic regurgitation as severe by correlating the records with the other usual indices | Day 1
  It allows tele-diastolic velocity measurement at the left subclavian artery
Establish a speed ratio threshold (systolic peak / tele-diastolic velocity) at the aortic arch and left subclavian artery | Day 1
  Diastolic / systolic speed ratio measurement at the left subclavian artery
Evaluate the appearance of distal anterior interventricular flow and analyze its association with the severity of aortic leakage | Day 1
  It allows to evaluate the changes in coronary flow morphology (diastolic / systolic velocity, and S / D ratio) in anterior interventricular during severe aortic regurgitation
Evaluate the 4D flow MRI parameters | Day 1
  It allows the measurement of regurgitant and anterograde volume in 4D flow MRI at the same sites as transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Olivier LOZINGUEZ, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided